CLINICAL TRIAL: NCT00265161
Title: The Effectiveness of Influenza Vaccine Among Health Care Workers in a Hospital Setting.
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Other Study IDs: 4180905
Record Dates: First submitted 2005-12-12; First posted 2005-12-14 (Estimated); Last update posted 2007-06-01 (Estimated); Status verified 2006-08

CONDITIONS: Influenza Vaccines
Keywords: influenza vaccine; effectiveness; health care worker; OBSERVATIONAL STUDY
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The study will be held in the winter of 2005-2007. The aim is to assess the effectiveness of the influenza vaccine in health care workers (HCW).

DETAILED DESCRIPTION:
The study will be held in the winter of 2005-2006. Groups of vaccinated HCW and not vaccinated HCW will be followed for symptoms suggestive of influenza. For each event a quick through test for influenza A or B will be done and if positive will be confirmed by viral study. Data regarding days of illness, absence from work, therapy etc., will be collected. Effectiveness will be calculated as well as cost/effectiveness of vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Previously healthy health care worker vaccinated or not

Exclusion Criteria:

* Immunocompromised state

Min Age: 18 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40
Dates: Start 2005-12; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Miron, MD, Principal Investigator — HaEmek Medicak Center, Afula, Israel
Locations (1):
- Pediatric Dpt A', HaEmek Medical Center, Afula, Israel